CLINICAL TRIAL: NCT04222361
Title: Prevention of Acute Renal Injury in the Septic Patient by Implementing the KDIGO Guideline in High-risk Patients Identified by Biomarkers
Brief Title: KDIGO Bundle to Prevent AKI in Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, María Mercader Alarcón, Principal Investigator, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI 42/2018
Record Dates: First submitted 2020-01-04; First posted 2020-01-10 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Septic Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KDIGO guide recommendations (Experimental): Preventive recommendations the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines for AKI
  Interventions: Procedure: Preventive recommendations for kidney disease: guidelines for improving overall outcomes (KDIGO) for AKI
- Standard care (No Intervention): The patients assigned to the control group will receive the current standard care of the septic patients of the Unit according to our protocols

INTERVENTIONS:
Procedure: Preventive recommendations for kidney disease: guidelines for improving overall outcomes (KDIGO) for AKI — Patients assigned to the treatment group will receive the AKI preventive recommendations from the KDIGO guide: withdraw nephrotoxics, ensure volemia and renal perfusion pressure by means of advanced hemodynamic monitoring-optimization (minimum monitoring objective: Unit algorithm based on volume systolic (VS) by pulse wave analysis - Flotrac® / ClearSight® system - or transpulmonary thermodilution - VolumeView® system -), monitor plasma creatinine and urinary expenditure, avoid hyperglycemia (serum blood glucose target: 110-149 mg / dl), and consider alternatives to diagnostic-therapeutic radiocontrast procedures.
  Arms: KDIGO guide recommendations

SUMMARY:
Summary: Controlled, prospective, randomized and randomized clinical trial of two intervention groups (standard care vs. preventive recommendations the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines for AKI) of patients diagnosed with sepsis and abdominal post-surgical septic shock with positive results in the risk determination of acute renal injury by NephroCheck® Test that integrates the urinary biomarkers TIMP-2 and IGFBP-7.

Hypothesis: The implementation of a package of preventive measures proposed by the KDIGO guide can reduce the occurrence and severity of acute renal injury in the high-risk abdominal post-surgical septic patient detected by urinary biomarkers for early detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients (or their informed family members) who accept and sign the informed consent.
* Patients diagnosed with sepsis or abdominal post-surgical septic shock.

Exclusion Criteria:

* Patients under 18 years.
* Patients (or their authorized relatives) who refuse to sign the informed consent.
* Patients diagnosed with sepsis or non-surgical septic shock.
* Patients diagnosed with sepsis or septic shock of origin other than abdominal.
* Patients with AKI stages KDIGO 2 and 3 and / or renal replacement therapy.
* Patients with chronic renal failure and glomerular filtration <30 ml / min and / or undergoing treatment with dialysis or previous renal transplantation.
* Patients with AKI of origin other than the diagnosed septic, such as glomerulonephritis or interstitial nephritis, renal artery occlusion and / or postrenal obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Compare the incidence of moderate-severe acute renal injury | 72 hours
  Compare the incidence of moderate-severe acute renal injury (stages KDIGO 2 and 3) in the first 72 hours of diagnosis of sepsis and septic post-surgical septic shock in patients at high risk of AKI determined by NephroCheck® Test (those with a ≥0.3 ng / ml2 / 1000 result) that the package of preventive measures proposed by the KDIGO guideline is applied vs. standard treatment

SECONDARY OUTCOMES:
Compare mortality from any cause | 90 days
  Compare mortality from any cause at 12, 24, 48 and 72 hours, and 30, 60 and 90 days in patients diagnosed with sepsis and abdominal post-surgical septic shock and high risk of AKI determined by NephroCheck® Test (patients with results ≥0.3 ng / ml2 / 1000) that the package of preventive measures proposed by the KDIGO guideline is applied vs. standard treatment
Compare the number of participants in need of renal replacement therapy | 90 days
  Compare the number of participants in need of renal replacement therapy at 12, 24, 48 and 72 hours, and 30, 60 and 90 days in patients diagnosed with sepsis and abdominal post-surgical septic shock and high risk of AKI determined by NephroCheck® Test (those with result ≥0.3 ng / ml2 / 1000) that the package of preventive measures proposed by the KDIGO guideline is applied vs. standard treatment
Compare the number of participants with persistent renal dysfunction | 90 days
  Compare the number of participants with persistent renal dysfunction at 30, 60 and 90 days in patients diagnosed with sepsis and abdominal post-surgical septic shock and high risk of AKI determined by NephroCheck® Test (those with a ≥0.3 ng / ml2 / 1000 result) that the package of preventive measures proposed by the KDIGO guideline is applied vs. standard treatment
Compare the number of days of stay in the Surgical ICU | 90 days
  Compare the number of days of stay in the Surgical ICU in patients diagnosed with sepsis and septic post-surgical septic shock and high risk of AKI determined by NephroCheck® Test (those with a result ≥0.3 ng / ml2 / 1000) that apply the package of preventive measures proposed by the guide KDIGO vs. standard treatment
Compare the number of days of stay in the hospital | 90 days
  Compare the number of days of stay in the hospital in patients diagnosed with sepsis and abdominal post-surgical septic shock and high risk of AKI determined by NephroCheck® Test (those with a result ≥0.3 ng / ml2 / 1000) that apply the package of preventive measures proposed by the KDIGO guide vs. standard treatment
Measure the incidence of development of AKI in patients at low risk of AKI determined by NephroCheck® Test | 72 hours
  Measure the incidence of development of AKI (any KDIGO stage) at 12, 24, 48 and 72 hours after diagnosis of sepsis and septic post-surgical septic shock in patients at low risk of AKI determined by NephroCheck® Test (those with a result of 0.3 ng / ml2 / 1000).

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Intensive Care Unit of the General University Hospital of Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No